CLINICAL TRIAL: NCT03670173
Title: Safety and Efficacy Assessments of Osalmid in the Treatment of Multiple Myeloma
Brief Title: Safety and Efficacy Assessments of Osalmid in Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Jumei Shi, Professor, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STPH-MM001
Record Dates: First submitted 2018-09-09; First posted 2018-09-13 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma, Osalmid
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: multi-center, single-arm, open-label, non-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osalmid (Experimental): Participants are initially given oral capsules with 0.5g tid osalmid daily for two weeks. Thereafter, the dosage will be increased by 0.25g tid every two weeks as tolerated by participants to a maximum daily dosage of 1.0g tid for up to one year. One course of osalmid treatment lasts four weeks. Response will be assessed at the end of each treatment course, and patients who have achieved MR (minor remission) or more than MR at the end of the fourth course will continue to take 1.0g tid osalmid daily for consolidation / maintenance therapy. Otherwise, patients who have not achieved MR at the end of the fourth course and patients who are assessed for PD (progression of disease) at the end of each course will receive salvage treatment, such as a combined treatment of osalmid and dexamethasone or the VCD (bortezomib, cyclophosphamide and dexamethasone) regimen.
  Interventions: Drug: Osalmid

INTERVENTIONS:
Drug: Osalmid — Participants are initially given oral capsules with 0.5g tid osalmid daily for two weeks. Thereafter, the dosage will be increased by 0.25g tid every two weeks as tolerated by participants to a maximum daily dosage of 1.0g tid for up to one year.
  Other Names: 2-hydroxy-N-(4-hydroxyphenyl)-benzamide

SUMMARY:
This study aims to evaluate the safety and efficacy of a traditional cholagogue drug osalmid, 2-hydroxy-N-(4-hydroxyphenyl)-benzamide, in the treatment of multiple myeloma (MM).

DETAILED DESCRIPTION:
Osalmid, 2-hydroxy-N-(4-hydroxyphenyl)-benzamide, is a traditional cholagogue and is clinically used in China to promote biliary drainage and protect liver function. Studies have shown that osalmid is an inhibitor of ribonucleotide reductase (RR). Recently, it was proven by our group that osalmid induced a dose-dependent lethality in multiple myeloma (MM) cell lines H929, OPM2, U266, OCI-MY5, and RPMI 8266, as well as in MM xenograft mouse models. This study aims to assess the safety and efficacy of osalmid in the treatment of MM.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age≥ 18 years old who are willing to receive the treatment of osalmid;
2. Patients must be diagnosed with active and measurable (symptomatic) multiple myeloma according to IMWG 2003/WHO 2008(V4) MM diagnosis criteria detailed as following:1). Positive M protein in serum and/or urine; 2). Pathologically diagnosed with multiple myeloma or found colonic plasma cells in bone marrow; 3). At least one symptom of related organ damage or tissue lesion: a. hypercalcemia: serum calcium increases 0.25mmol/L or more over upper limit of normal value(ULN) or > 2.75mmol/L; b. anemia: Hemoglobin decreases 20g/L or more over lower limit of normal value(LLN) or <100g/L；c. bone lesion: lytic bone lesion or osteoporosis accompanied with compressive fracture (confirmed with MRI、CT or PET-CT); d. others: symptomatic hyperviscosity, amyloidosis, recurrent infection (more than twice within 12 months);
3. Eastern Cancer Organization Group (ECOG) score≤2 and expected survival>2 months;
4. Belongs to "measurable disease": serum M protein ≥10g/L and/or 24 hour urine M protein ≥200mg;
5. No active infectious diseases;
6. No severe organic dysfunction (except renal function insufficiency caused by multiple myeloma), lab results must meet the following criteria (within 7 days before initiation of therapy): a. Total bilirubin ≤ 1.5*ULN (same age group); b. AST and ALT ≤ 2.5*ULN (same age group); c. Cardiac enzyme < 2*ULN (same age group); d. Normal ejection fraction confirmed in echo;
7. Able to swallow oral medicine;
8. Volunteer to participate into this clinical trial and the informed consents must be written by patients themselves or their direct relatives. Authorized medical attorney or direct relatives can write the informed consents if it is not good for patients' treatment when consider the severity of their disease.

Exclusion Criteria:

1. Received anti-myeloma treatment before (not include radiotherapy, bisphosphonates or single short term steroids treatment [the dose and duration of prednisone should be no more than 40mg/d and 4 days and should discontinue this treatment within 14 days before the enrollment]);
2. Primary or secondary plasma cell leukemia;
3. Positive HIV tests or active infection phase of HAV, HBV and HCV; or HBV DNA copies >104/ml；AST and ALT > 2.5*ULN (same age group);
4. Severe diseases that threaten patients with unacceptable risks; these diseases include but are not confined to unstable heart diseases, which can be defined as cardiac accidents such as MI within 6 months, NYHA stage Ⅲ-Ⅳ heart failure, uncontrolled atrial fibrillation or hypertension and myeloma requiring long term administration of steroids or immune-inhibitors;
5. Renal failure requiring hemodialysis or peritoneal dialysis;
6. Severe embolic or thrombotic events before therapy;
7. Major surgery within 30 days before being enrolled;
8. Total obstruction of biliary tract;
9. Glaucoma;
10. History of malignancies except multiple myeloma unless being cured for more than 3 years;
11. Severe allergic to osalmide capsule;
12. Gestation, lactation or disagreed pregnancy;
13. Severe infectious diseases (uncured tuberculosis, pulmonary aspergillosis);
14. Seizures requiring medicines, patients with dementias and other mental disorders who cannot understand or obey the protocol;
15. Substance abuse, medical, psychological, or social conditions that may interfere with the subject's compliance in the study or assessment of the results of the study;
16. Severe liver and kidney dysfunction;
17. Patients who are considered unsuitable for enrollment by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-05-18 (Estimated); Study Completion 2021-05-18 (Estimated)

PRIMARY OUTCOMES:
overall response rate | at week16
  M protein qualification in serum and/or urine decline of at least 25%, 50%, 75%, or 90%

SECONDARY OUTCOMES:
time to progression | at week 48
  from the start of therapy to disease progression
duration of response | at week 48
  from the time response was achieved to disease progression or death
progression-free survival | at week 48
  from study entry to disease progression or death
overall survival | at week 48
  from the date of study entry to the date of death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jumei Shi, MD PhD, Study Director — Shanghai 10th People's Hospital; Weiliang Zhu, PhD, Principal Investigator — Shanghai Institute of Materia Medica, Chinese Academy of Sciences
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah N, Callander N, Ganguly S, Gul Z, Hamadani M, Costa L, Sengsayadeth S, Abidi M, Hari P, Mohty M, Chen YB, Koreth J, Landau H, Lazarus H, Leather H, Majhail N, Nath R, Osman K, Perales MA, Schriber J, Shaughnessy P, Vesole D, Vij R, Wingard J, Giralt S, Savani BN; American Society for Blood and Marrow Transplantation. Hematopoietic Stem Cell Transplantation for Multiple Myeloma: Guidelines from the American Society for Blood and Marrow Transplantation. Biol Blood Marrow Transplant. 2015 Jul;21(7):1155-66. doi: 10.1016/j.bbmt.2015.03.002. Epub 2015 Mar 11. PMID 25769794
- [Background] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696
- [Background] Rajkumar SV, Blood E, Vesole D, Fonseca R, Greipp PR; Eastern Cooperative Oncology Group. Phase III clinical trial of thalidomide plus dexamethasone compared with dexamethasone alone in newly diagnosed multiple myeloma: a clinical trial coordinated by the Eastern Cooperative Oncology Group. J Clin Oncol. 2006 Jan 20;24(3):431-6. doi: 10.1200/JCO.2005.03.0221. Epub 2005 Dec 19. PMID 16365178
- [Background] Rajkumar SV, Rosinol L, Hussein M, Catalano J, Jedrzejczak W, Lucy L, Olesnyckyj M, Yu Z, Knight R, Zeldis JB, Blade J. Multicenter, randomized, double-blind, placebo-controlled study of thalidomide plus dexamethasone compared with dexamethasone as initial therapy for newly diagnosed multiple myeloma. J Clin Oncol. 2008 May 1;26(13):2171-7. doi: 10.1200/JCO.2007.14.1853. Epub 2008 Mar 24. PMID 18362366
- [Background] Murakami H, Handa H, Abe M, Iida S, Ishii A, Ishikawa T, Ishida T, Oota M, Ozaki S, Kosaka M, Sakai A, Sawamura M, Shimazaki C, Shimizu K, Takagi T, Hata H, Fukuhara T, Fujii H, Miyata A, Wakayama T, Takatsuki K. Low-dose thalidomide plus low-dose dexamethasone therapy in patients with refractory multiple myeloma. Eur J Haematol. 2007 Sep;79(3):234-9. doi: 10.1111/j.1600-0609.2007.00908.x. Epub 2007 Jul 26. PMID 17655699
- [Background] Cavo M, Zamagni E, Tosi P, Tacchetti P, Cellini C, Cangini D, de Vivo A, Testoni N, Nicci C, Terragna C, Grafone T, Perrone G, Ceccolini M, Tura S, Baccarani M; Bologna 2002 study. Superiority of thalidomide and dexamethasone over vincristine-doxorubicindexamethasone (VAD) as primary therapy in preparation for autologous transplantation for multiple myeloma. Blood. 2005 Jul 1;106(1):35-9. doi: 10.1182/blood-2005-02-0522. Epub 2005 Mar 10. PMID 15761019
- [Background] Mikhael JR, Dingli D, Roy V, Reeder CB, Buadi FK, Hayman SR, Dispenzieri A, Fonseca R, Sher T, Kyle RA, Lin Y, Russell SJ, Kumar S, Bergsagel PL, Zeldenrust SR, Leung N, Drake MT, Kapoor P, Ansell SM, Witzig TE, Lust JA, Dalton RJ, Gertz MA, Stewart AK, Rajkumar SV, Chanan-Khan A, Lacy MQ; Mayo Clinic. Management of newly diagnosed symptomatic multiple myeloma: updated Mayo Stratification of Myeloma and Risk-Adapted Therapy (mSMART) consensus guidelines 2013. Mayo Clin Proc. 2013 Apr;88(4):360-76. doi: 10.1016/j.mayocp.2013.01.019. PMID 23541011
- [Background] Kyle RA, Rajkumar SV. Criteria for diagnosis, staging, risk stratification and response assessment of multiple myeloma. Leukemia. 2009 Jan;23(1):3-9. doi: 10.1038/leu.2008.291. Epub 2008 Oct 30. PMID 18971951
- [Background] Kapoor P, Fonseca R, Rajkumar SV, Sinha S, Gertz MA, Stewart AK, Bergsagel PL, Lacy MQ, Dingli DD, Ketterling RP, Buadi F, Kyle RA, Witzig TE, Greipp PR, Dispenzieri A, Kumar S. Evidence for cytogenetic and fluorescence in situ hybridization risk stratification of newly diagnosed multiple myeloma in the era of novel therapie. Mayo Clin Proc. 2010 Jun;85(6):532-7. doi: 10.4065/mcp.2009.0677. PMID 20511484
- [Background] Rajkumar SV. Updated Diagnostic Criteria and Staging System for Multiple Myeloma. Am Soc Clin Oncol Educ Book. 2016;35:e418-23. doi: 10.1200/EDBK_159009. PMID 27249749
- [Background] Rajkumar SV, Harousseau JL, Durie B, Anderson KC, Dimopoulos M, Kyle R, Blade J, Richardson P, Orlowski R, Siegel D, Jagannath S, Facon T, Avet-Loiseau H, Lonial S, Palumbo A, Zonder J, Ludwig H, Vesole D, Sezer O, Munshi NC, San Miguel J; International Myeloma Workshop Consensus Panel 1. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011 May 5;117(18):4691-5. doi: 10.1182/blood-2010-10-299487. Epub 2011 Feb 3. PMID 21292775
- [Derived] Xie Y, Wang Y, Xu Z, Lu Y, Song D, Gao L, Yu D, Li B, Chen G, Zhang H, Feng Q, Zhang Y, Hu K, Huang C, Peng Y, Wu X, Mao Z, Shao J, Zhu W, Shi J. Preclinical validation and phase I trial of 4-hydroxysalicylanilide, targeting ribonucleotide reductase mediated dNTP synthesis in multiple myeloma. J Biomed Sci. 2022 May 12;29(1):32. doi: 10.1186/s12929-022-00813-2. PMID 35546402